CLINICAL TRIAL: NCT05015023
Title: Effectiveness of Health Education Provided to Couples on Knowledge, Attitude, and Utilization of Maternity Waiting Homes in Hadiya Zone, Southern Ethiopia: A Cluster-Randomized Controlled Trial
Brief Title: Effectiveness of Health Education Provided to Couples on Utilization of Maternity Waiting Homes in Rural Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Teklemariam Yarinbab, MPH, Assistant Professor, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RP0901/11
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Maternal Death; Maternal Behavior
Keywords: maternity waiting home, male partner, Ethiopia
MeSH Terms: conditions — Maternal Death | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: The study will have two arms, i.e., intervention and control groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The behavioral intervention will be conducted on the experimental group for consecutive six months. The components of the intervention will be group health education, provision of IEC materials/Leaflets, and home visits.
  Interventions: Behavioral: Behavioral intervention
- Control (No Intervention): The routine care will be continued in the control group.

INTERVENTIONS:
Behavioral: Behavioral intervention — A cluster-randomized controlled trial will be conducted.
  Arms: Intervention

SUMMARY:
Maternity waiting homes (MWHs) were identified as a solution to improve pregnancy outcomes by bringing women living in geographically isolated areas closer to a healthcare facility. Literature shows that MWHs contribute significantly to the reduction of maternal death and stillbirth among users. Despite its importance in improving maternal & neonatal health outcomes, the utilization of MWHs is very low in Ethiopia. It is important to investigate what strategies could be effective in improving MWH utilization. Therefore, in this study cluster-randomized controlled trials will be conducted to evaluate the effect of male partner involvement intervention on MWH utilization in Ethiopia.

DETAILED DESCRIPTION:
The primary cause of adverse maternal health outcomes has been identified to be the delay in reaching care. This is often attributed to the long distances women need to travel to gain access to health facilities. Literature shows that maternity waiting homes contribute significantly to the reduction of maternal death and stillbirth among users. Despite its importance in improving maternal and neonatal health outcomes, the utilization of MWHs is very low in Ethiopia. So, it is important to investigate what strategies could be effective in improving MWH utilization in Ethiopia.

The aim of this study is to evaluate the effect of male partner involvement intervention on MWH utilization in Hadiya Zone, Southern Ethiopia. A cluster-randomized controlled trial will be performed. The intervention will have two arms, i.e., intervention and control. It will be a behavioral intervention. The interventions will be health education, home visit, and the provision of Information Education Communication (IEC) materials/leaflets. Health education will be delivered to "husband-expectant wife" pairs at the baseline. Then home visits will be conducted two times (in the third and fifth months of the intervention period). Leaflets will be provided to the study participants three times, i.e., at the baseline and during every home visit. The study participants will be pregnant women at the beginning of their second trimester living with their male partners at the time of the study.

Randomization will be conducted at the cluster level. Clusters will be Kebeles'. There will be 16 clusters or Kebeles. Data collectors (assessors) will be masked. The trial sample size will be 320 [160 in each arm]. A Generalized Estimating Equations model will be used. Data analysis will be conducted by SPSS or STATA software (as appropriate) using an Intention-To-Treat Approach. The duration of the intervention will be six months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at the beginning of second trimesters (14-16 weeks of gestation)
* Pregnant women currently live with their male partners
* Pregnant women permanent residents of the study area
* Pregnant women live in a place ≥2 hours of walking distance from the nearest health facility and/or have no access to public transportation
* Pregnant women whose husbands/male partners will be willing to participate in the study

Exclusion Criteria:

* Pregnant women ≤ 13 weeks of gestation
* Pregnant women not living with their male partners at the time of the study
* Pregnant women who are not permanent residents of the study area
* Pregnant women live in a place < 2 hours of walking distance from the nearest health facility or have access to transportation
* Pregnant women whose husbands are not willing to participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Utilization of MWH | up to six months
  Utilization of MWH is the use of MWHs by pregnant women in their final weeks of pregnancy to bridge the geographic gap in obstetric care. It is the proportion of pregnant women who use MWHs in the final weeks of pregnancy among the eligible women who are study participants.

SECONDARY OUTCOMES:
Level of Maternal Knowledge and Attitude | up to six months
  Knowledge will be measured using 'Yes' or 'No' questions and attitude will be measured using the Likert scale. There will be 7 questions for the knowledge assessment and 5 questions with 5 points Likert scales for the attitude assessment. Individual scores on each item will be added to yield the sum score. Participants who score above the median in the assessment will be regarded to be knowledgeable or have a good attitude about MWHs, while those who score below the median will be judged to have poor knowledge or an unfavorable attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Teklemariam E Yarinbab, MPH, Principal Investigator — Mizan Tepi University; Hailay A Gesesew, PhD, Principal Investigator — Torrens University Australia; Tefera Belachew, PhD, Principal Investigator — Jimma University
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Derived] Yarinbab TE, Gesesew HA, Belachew T. Effect of health education provided to couples on maternal knowledge, attitude and use of maternity waiting homes in rural Ethiopia: A cluster-randomized trial. Midwifery. 2024 Nov;138:104153. doi: 10.1016/j.midw.2024.104153. Epub 2024 Aug 22. PMID 39197275
- [Derived] Yarinbab TE, Gesesew HA, Harrison MS, Belachew T. Effect of couple-based health education on male-partners knowledge and attitude towards maternity waiting homes in rural Ethiopia: a cluster-randomized trial. Sci Rep. 2023 Oct 27;13(1):18446. doi: 10.1038/s41598-023-45681-4. PMID 37891206